CLINICAL TRIAL: NCT00500578
Title: A Randomized Study Evaluating Two Different Schedules of Aerosolized Ribavirin For Treatment of RSV Upper Respiratory Infections in Patients With Hematological Malignancies
Brief Title: Intermittent Use of Aerosolized Ribavirin for Treatment of RSV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: ICN Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID03-0010
Record Dates: First submitted 2007-07-10; First posted 2007-07-12 (Estimated); Results first posted 2010-09-16 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Hematological Malignancies
Keywords: Hematological Malignancies; Respiratory Infection; Respiratory Syncytial Virus; RSV; Ribavirin; Virazole
MeSH Terms: conditions — Hematologic Neoplasms; Respiratory Tract Infections | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: Standard Schedule - Ribavirin (Experimental): Aerosolized Ribavirin 6 grams over 18 hours every 24 hours
  Interventions: Drug: Ribavirin
- 2: Modified Schedule - Ribavirin (Experimental): Aerosolized Ribavirin 2 grams over 3 hours every 8 hours
  Interventions: Drug: Ribavirin

INTERVENTIONS:
Drug: Ribavirin — Arm 1 = 6 Grams Over 18 hours Every 24 Hours
  Other Names: Virazole
  Arms: 1: Standard Schedule - Ribavirin
Drug: Ribavirin — Arm 2 = 2 Grams Over 3 Hours Every 8 Hours.
  Other Names: Virazole
  Arms: 2: Modified Schedule - Ribavirin

SUMMARY:
Primary Objectives:

1. To determine whether aerosolized ribavirin is effective when given at an intermittent dose over 3 hours every 8 hours for therapy of RSV upper respiratory tract infection (URI) and whether it can prevent progression to pneumonia.
2. To determine the effect of this regimen on persistence of viral shedding.

DETAILED DESCRIPTION:
Ribavirin is the drug that is normally given to treat upper respiratory infections caused by RSV. The drug is only effective when inhaled as an aerosol. This treatment requires the patient to be in a tent and inhale the medication. The usual method for administering this drug has been to inhale the medication continuously over 18 hours. In this study, the same total dose of the medication will be used, however, treatment will be for 3 hours every 8 hours.

As part of your standard care, before treatment you will have blood drawn (around 2 teaspoons) for routine blood tests. You will have a washing from your throat and nose collected. For this procedure, around 1 teaspoon of saline will be sprayed into each nostril and you will blow your nose into a cup. You will have a swab of the nose and throat. You will also have a chest x-ray to check on the status of the disease. Women who are able to have children must have a negative blood or urine pregnancy test.

Before treatment, you will be randomly assigned (as in the toss of a coin) to one of two groups. Participants in one group will receive treatment with ribavirin over 3 hours every 8 hours. Participants in the other group will receive treatment using the standard treatment schedule, ribavirin over 18 hours every 24 hours.

For both groups, the drug will be administered as an aerosol using a face mask. This will require you to be in a tent while you are receiving therapy. Treatment will last between 5 and 10 days. This will require hospitalization. In addition to ribavirin treatment, you will also receive Xopenex inhalation therapy every 6 - 8 hours. Xopenex is a drug designed to make breathing easier. We may need to use another breathing treatment, albuterol inhalation therapy for one time if needed, directly after receiving ribavirin to make breathing easier.

Every 2-4 days during treatment you will have blood collected (around 2 teaspoons) for routine tests. On Days 3 and 7 of treatment (+/- 2 days), you will have a repeat throat and nose washings/swabs. The washings and swabs will then be repeated once a week for 2 weeks, or until 2 consecutive cultures are negative, if that occurs sooner. If your doctor feels it is necessary, you may have a repeat chest x-ray.

If at any time you develop signs of pneumonia, you will be removed from the study and will be treated with the standard schedule of ribavirin by continuous inhalation and/or other therapy for 18 hours a day. Also, if you develop any intolerable side effects, you will be taken off the study and your doctor will discuss other treatment options with you.

This is an investigational study. Ribavirin is FDA approved and is commercially available. However, the method of administration of ribavirin is investigational. Up to 50 patients will participate in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with these underlying malignancies will be eligible for this study: Autologous BMT patients, Allogeneic BMT patients, and patients with hematological malignancy.
2. Patients must be at least 5 years of age.
3. Only patients with infection limited to the URT will be eligible for entry on study
4. Patients will be eligible for entry on study if a nasopharyngeal wash or throat swab specimen is positive by rapid RSV antigen testing or by a positive culture for RSV.

Exclusion Criteria:

1. Patients with evidence of RSV LRTI as documented by a positive rapid RSV antigen testing or by a positive culture for RSV from a nasopharyngeal wash or throat swab AND new infiltrates on chest radiograph and/or abnormal blood gas determination
2. Patients with hypersensitivity to ribavirin or its components
3. Pregnant women. Participants must practice birth control during the study if they are sexually active. If the participant is pregnant, she may not be enrolled on this study. Mothers should refrain from breast-feeding during the study to avoid injury to their children.
4. Patients with positive RSV by rapid testing or culture in bronchoalveolar lavage regardless of the chest radiographic results.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2003-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy F. Chemaly, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Chemaly RF, Torres HA, Munsell MF, Shah DP, Rathod DB, Bodey GP, Hosing C, Saifan C, Raad II, Champlin RE. An adaptive randomized trial of an intermittent dosing schedule of aerosolized ribavirin in patients with cancer and respiratory syncytial virus infection. J Infect Dis. 2012 Nov;206(9):1367-71. doi: 10.1093/infdis/jis516. Epub 2012 Aug 22. PMID 22927454
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty patients were enrolled between October 2003 and March 2008, either from the outpatient settings or inpatients. Eligible patients were randomized to either Arm 1 (Standard regimen: 6gm over 18 hours every 24 hours) or Arm 2 (Modified regimen: 6gm over 3 hours every 8 hours).
Pre-assignment Details: Only one patient was excluded from the trial after enrollment and before starting the intervention because his Chest X-Ray was read later on as positive for infiltrates.
Groups:
- Standard Schedule - Ribavarin: Aerosolized Ribavirin 6 gm over 18 hours every 24 hours
- Modified Schedule - Ribavarin: Aerosolized Ribavirin 6 gm over 3 hours every 8 hours
Period: Overall Study
Arm/Group | Standard Schedule - Ribavarin | Modified Schedule - Ribavarin
Started | 18 | 32
Completed | 18 (All completed) | 32 (All completed)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Schedule - Ribavarin | Modified Schedule - Ribavarin | Total
Number analyzed (Participants) | 18 | 32 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 17 | 27 | 44
  >=65 years | 1 | 4 | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 47.9 (11.44) | 46.7 (14.35) | 47.16 (13.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 21
  Male | 9 | 20 | 29
Region of Enrollment [Number; unit: participants]
  United States | 18 | 32 | 50

OUTCOME MEASURES:

1. Primary Outcome: Occurrences of Pneumonia
Description: Treatment failure defined as progression to pneumonia within 7 days of initial treatment with aerosolized ribavirin. Patients considered as a failure or to have an unfavorable response if there develop signs and symptoms of pneumonia during therapy either evidenced by chest-xray or clinically, meaning they did reach the primary endpoint.
Time Frame: 6 Years
Population: The analysis was carried out per protocol. All patients enrolled were included in the final analysis except one patient who was a screen failure.
Measure: Number; unit: Participants
Arm/Group | Standard Schedule - Ribavarin | Modified Schedule - Ribavarin
Number analyzed (Participants) | 18 | 32
Participants | 4 | 3

ADVERSE EVENTS:
Time Frame: 6 Years
Arm/Group | Standard Schedule - Ribavarin | Modified Schedule - Ribavarin
Serious Adverse Events (participants affected / at risk) | 2/18 | 4/32
Other Adverse Events (participants affected / at risk) | 0/18 | 0/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Schedule - Ribavarin (N=18) | Modified Schedule - Ribavarin (N=32)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 4 (6) — Severe diarrhea occured in 1 patient
Bladder Spasm (Renal and urinary disorders) | 0 (0) | 1 (1) — Occured in 1 patient
Acute Graft Versus Host Disease (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Affected 1 patient
Chronic Graft Versus Host Disease (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Affected 1 patient
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Occured in 1 patient
Anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Elevated creatinine (Renal and urinary disorders) | 0 (0) | 1 (1)
Hyperglycemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Elevated Transaminase Level (Hepatobiliary disorders) | 1 (1) | 0 (0)
Elevated Bilirubin level (Hepatobiliary disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The interpretation of our data is limited by our study's open-label design, which may bias assessments of tolerability or toxicity but would be less likely to bias assessments of therapeutic endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No